CLINICAL TRIAL: NCT03240601
Title: Combined Influence of Transcutaneous Spinal Cord Stimulation and Locomotor Training on Spasticity and Walking Outcomes After Spinal Cord Injury
Brief Title: Spinal Cord Stimulation to Augment Activity Based Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shepherd Center, Atlanta GA (Other)
Collaborators: Foundation Wings For Life (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 696
Record Dates: First submitted 2017-07-17; First posted 2017-08-07 (Actual); Results first posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2021-12

CONDITIONS: Transcutaneous Spinal Stimulation; Walking; Spasticity; Human; Spinal Cord Injuries
MeSH Terms: conditions — Muscle Spasticity; Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Subthreshold (Sham Comparator): Individuals will undergo their standard physical therapist directed locomotor training while receiving transcutaneous spinal cord stimulation. The stimulation intensity will briefly ramp up to the lowest intensity that is first detected by the participant and then ramped down to a level no longer detected by the participant. Participants will continue their locomotor training.
  Interventions: Device: Transcutaneous spinal stimulation
- Active (Experimental): Individuals will undergo their standard physical therapist directed locomotor training while receiving transcutaneous spinal cord stimulation. The stimulation intensity will ramp up slowly to a level that produces parasthesia (tingling) throughout the lower extremity. This intensity will be applied for 30 minutes while participants continue their locomotor training.
  Interventions: Device: Transcutaneous spinal stimulation

INTERVENTIONS:
Device: Transcutaneous spinal stimulation — For TSS, a transcutaneous electrical nerve stimulation (TENS) unit is used. A 2 inch diameter round electrode is placed on the skin over T11/T12 (cathode), and a large butterfly electrode is placed on the skin over the umbilicus (anode). Pulse width is set to 400 microseconds at 50 Hz.
  Other Names: TSS

SUMMARY:
Involuntary muscle activity, often called spasticity, is a common problem following spinal cord injury (SCI) that can make it hard to move. Many things can cause spasticity including: muscle stretch, movement, or it can happen for no reason, and it is often described as an uncontrolled muscle spasm or feeling of stiffness. Drugs are typically used to treat spasticity, but they often have side effects, like muscle weakness, which can add to movement problems. Rehabilitation therapies offer alternatives to drugs for treating involuntary muscle activity, and rehabilitation can also improve daily function and quality of life. These benefits may be greater when several rehabilitation therapies are used together.

Walking ability can be improved with a type of therapy called "locomotor training". This type of therapy may also have the benefit of decreasing spasticity. When locomotor training (LT) is combined with electrical stimulation, the benefits of training may be increased. In this study, investigators will use a kind of stimulation called transcutaneous spinal cord stimulation ("TSS") to stimulate participants' spinal cord nerves during locomotor training.

DETAILED DESCRIPTION:
Involuntary muscle activity, often referred to as spasticity, is a common problem following spinal cord injury. Spasticity can be evoked by stimuli or occur spontaneously, and it can manifest as spasms, clonus, or the stiffness associated with hypertonia. While medications are typically used to treat the general symptoms of spasticity, they often have additional side effects, like muscle weakness, that can impede rehabilitation. Physical therapeutics offer an alternative to these drug treatments, but the most effective therapeutic strategy for managing spasticity has not yet been identified. A combination of physical therapeutics may provide the best strategy for managing spasticity while also improving general motor control for functional movements.

Walking ability can be improved through locomotor training, which has also been shown to reduce spasticity. When locomotor training is combined with electrical stimulation, the benefits of training may be increased. To investigate the potential benefits of this combinatorial treatment strategy, investigators will use a kind of electrical stimulation called transcutaneous spinal cord stimulation ("TSS") to stimulate spinal cord nerves during locomotor training.

In order to facilitate the translation of study findings into clinical practice, this study uses a pragmatic design, meaning that the study will involve the use of real world clinical settings and practices. Participants will undergo their standard physical therapist directed locomotor training program while receiving transcutaneous spinal cord stimulation (TSS) as an additional treatment. The effects of locomotor training alone will be compared to the combination of locomotor training with TSS, specifically comparing the effects of these treatments on spasticity and walking function.

Investigators expect that the combination of TSS with locomotor training will provide 1) a greater reduction in spasticity and 2) a greater improvement of walking function compared to locomotor training alone.

The findings from this study have the potential to rapidly facilitate the translation of a novel combination treatment for the management of spasticity and improvement of walking function into real world clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to consent and/or authorize use of protected health information
* Be between 18-65 years of age
* Be enrolled in Spinal Cord Injury In-Patient or Day Program at the Shepherd Center
* Be eligible for locomotor training at the Shepherd Center
* Be able to take a step, with or without an assistive device
* Have a spinal cord injury, completed in-patient rehabilitation, and have been discharged to home
* Have at least mild "spasticity" affecting leg muscles
* You may participate if you use prescription medications, including baclofen for control of spasticity

Exclusion Criteria:

* Inability or unwillingness to consent and/or authorization for use of protected health information
* Progressive or potentially progressive spinal lesions, including degenerative, or progressive vascular disorders of the spine and/or spinal cord
* Neurologic level at or below spinal level T12
* History of cardiovascular irregularities
* Problems with following instructions
* Orthopedic problems that would limit your participation in the protocol (e.g. knee or hip flexion contractures of greater than 10 degrees)
* Women who are pregnant, or who have reason to believe they are or may become pregnant due to unknown risks to the fetus associated with tcSCS
* Persons who have implanted stimulators/electronic devices of any type will be excluded due to unknown potential of tcSCS effects
* Active infection of any type, as infection may exacerbate spasticity resulting in inability to identify the influence of the treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edelle C Field-Fote, PT, PhD, Principal Investigator — Shepherd Center, Inc
Locations (1):
- Shepherd Center, Inc., Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Subthreshold: Individuals will undergo their standard physical therapist directed locomotor training while receiving transcutaneous spinal cord stimulation. The stimulation intensity will briefly ramp up to the lowest intensity that is first detected by the participant and then ramped down to a level no longer detected by the participant. Participants will continue their locomotor training.
  Transcutaneous spinal cord stimulation: For tcSCS, a transcutaneous electrical nerve stimulation (TENS) unit is used. A 2 inch diameter round electrode is placed on the skin over T11/T12 (cathode), and a large butterfly electrode is placed on the skin over the umbilicus (anode). Pulse width is set to 400 microseconds at 50 Hz.
- Active: Individuals will undergo their standard physical therapist directed locomotor training while receiving transcutaneous spinal cord stimulation. The stimulation intensity will ramp up slowly to a level that produces parasthesia (tingling) throughout the lower extremity. This intensity will be applied for 30 minutes while participants continue their locomotor training.
  Transcutaneous spinal cord stimulation: For tcSCS, a transcutaneous electrical nerve stimulation (TENS) unit is used. A 2 inch diameter round electrode is placed on the skin over T11/T12 (cathode), and a large butterfly electrode is placed on the skin over the umbilicus (anode). Pulse width is set to 400 microseconds at 50 Hz.
Period: Overall Study
Arm/Group | Subthreshold | Active
Started | 9 | 9
Completed | 8 | 8
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subthreshold | Active | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 4 | 6 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Walking Function - 10m Walk Walking Speed (m/s)
Description: You will walk over a mat that contains sensors to measure your walking speed as well as wear motion tracking sensors. You will be allowed to use whatever assistive devices you typically use (e.g., braces, walker, forearm crutches). In addition to walking speed, we will also assess your gait kinematics.
Time Frame: Change in 10m Walk Speed (m/s) during the Intervention Phase (Week 2 test to Week 4 test)
Measure: Mean (Standard Deviation); unit: speed difference in meters per second
Arm/Group | Subthreshold | Active
Number analyzed (Participants) | 8 | 8
speed difference in meters per second | 0.06 (0.08) | 0.16 (0.13)

2. Primary Outcome: Change in Spasticity - Pendulum Test
Description: This test measures the amount of spasticity in your leg muscles. You will sit at the edge of a mat with your lower legs hanging over the edge of the mat. Motion capture sensors (Xsens) will be placed on both of your legs to record changes in your knee joint angles when your leg is dropped. The examiner will straighten your leg and then allow it to drop and swing over the edge of the mat. The angle of your knee and the movement of your leg will be recorded as it drops. This will be performed three times for each leg separately.
Time Frame: Pendulum angle (degrees) change during the Intervention Phase (Week 2 test to Week 4 test)
Measure: Mean (Standard Deviation); unit: Change in Angle (degrees)
Arm/Group | Subthreshold | Active
Number analyzed (Participants) | 8 | 8
Change in Angle (degrees) | 7 (13) | 7 (19)

3. Secondary Outcome: Change in Walking Function - 2 Minute Walk
Description: You will walk for 2 minutes overground and we will measure how far you walk.
Time Frame: 2 Minute Walk test (distance) change during the Intervention Phase (Week 2 test to Week 4 test)
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Subthreshold | Active
Number analyzed (Participants) | 8 | 8
meters | 7 (.03) | 15 (.12)

4. Secondary Outcome: Change in Spasticity - Ankle Clonus Drop Test
Description: This test measures the amount of spasticity in your ankle. We will use the motion capture sensors to record your ankle joint angles. For this test you will sit upright. Your leg will be raised to 10cm above the rest position and released allowing the front of your foot to land on the edge of a box. The angle bouncing movement of your foot (clonus) will be recorded as it drops and catches on the box. This will be performed three times for each leg separately. Full details of test methods can be found at: Manella, Roach, and Field-Fote. Temporal Indices of Ankle Clonus and Relationship to Electrophysiologic and Clinical Measures in Persons With Spinal Cord Injury. J Neurol Phys Ther. 2017 Oct;41(4):229-238.
Time Frame: Change in number of clonic ankle oscillations elicited via Ankle Clonus Drop Test during the Intervention Phase (Week 2 test to Week 4 test)
Measure: Mean (Standard Deviation); unit: change in clonic oscillations
Arm/Group | Subthreshold | Active
Number analyzed (Participants) | 8 | 8
change in clonic oscillations | 1 (7) | 1 (4)

5. Secondary Outcome: Change in Spasticity - Muscle Co-contraction During Voluntary Activation
Description: Muscle activity will be recorded using electromyography (EMG) during activities where you move your legs, and activities where your legs are moved by the examiner. Electrodes will be placed on four muscles of your legs (front and back of your thigh and lower leg), you will be asked to move your ankles and extend your legs while we record your muscle activity. We will test whether the EMG is activated in only one muscle (isolated) when you try to activate that muscle, or whether muscles that you are not trying to activate are also activated at the same time (co-contraction)
Time Frame: Co-contraction change during the Intervention Phase (Week 2 test to Week 4 test)
Measure: Mean (Standard Deviation); unit: change in co-contraction ratio
Arm/Group | Subthreshold | Active
Number analyzed (Participants) | 8 | 8
change in co-contraction ratio | 1 (3) | 1 (3)

6. Secondary Outcome: Change in Spasticity - Spinal Cord Assessment Tool for Spastic Reflexes (SCATS) Test
Description: A trained therapist will perform the SCATS assessment before and after each training session. SCATS assesses 3 aspects of spasticity: clonus, flexor spasms, extensor spasms in response to perturbation. Scores range from 0-3 as follows: 0 = no reaction; 1 = mild, <3 sec response; 2 = moderate, 3-10 sec response; 3 = severe, >10 sec response
Time Frame: SCATS scores change during the Intervention Phase (Week 2 test to Week 4 test)
Measure: Mean (Standard Deviation); unit: change in SCI-SET score
Arm/Group | Subthreshold | Active
Number analyzed (Participants) | 8 | 8
change in SCI-SET score | 0 (2) | 0 (2)

7. Secondary Outcome: Stimulation Tolerability
Description: Using a 0-10 numerical rating scale (NRS) for pain, you will be asked your perception of pain during the final 2 weeks of stimulation. NRS anchors are 0 = no pain, 10 = pain as bad as you can imagine
Time Frame: Numerical rating scale of painfulness of stimulation in stimulation group only during stimulation weeks only (weeks 3 and 4)
Population: Only the LT+TSS group received active stimulation, tolerability was assessed only in this group
Measure: Mean (Standard Deviation); unit: Scores on a 1-10 scale
Arm/Group | Subthreshold | Active
Number analyzed (Participants) | 0 | 8
Scores on a 1-10 scale |  | 3 (1)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Subthreshold | Active
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-28): https://cdn.clinicaltrials.gov/large-docs/01/NCT03240601/Prot_SAP_002.pdf